CLINICAL TRIAL: NCT04878549
Title: A Multisite Evaluation of Functional Genomic Signatures for the Improved Diagnosis of Acute Undifferentiated Febrile Infections
Brief Title: Transcriptomic Responses for the Identification of Pathogens
Acronym: TRiP
Status: Recruiting | Type: Observational
Sponsor: University of Sheffield (Other)
Collaborators: Christian Medical College, Vellore, India (Other); KEMRI-Wellcome Trust Collaborative Research Program (Other)
Responsible Party: Sponsor
Other Study IDs: 157365
Record Dates: First submitted 2021-01-20; First posted 2021-05-07 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Enteric Fever; Acute Febrile Illness; Typhoid; Paratyphoid Fever; Fever
Keywords: Gene Expression Profiling; RNA-Seq
MeSH Terms: conditions — Typhoid Fever; Paratyphoid Fever; Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Febrile Adults: 1200 adult participants (15 to 65 years old) with a febrile illness without localising features and reported duration of 3-14 days.
  Interventions: Diagnostic Test: 5-gene transcription signature
- Controls: 400 afebrile, healthy adult participants (15 to 65 years old).
  Interventions: Diagnostic Test: 5-gene transcription signature
- Febrile Children: 400 child participants (2 to 14 years old) with a febrile illness without localising features and reported duration of 3-14 days. This is an exploratory arm of the study.
  Interventions: Diagnostic Test: 5-gene transcription signature

INTERVENTIONS:
Diagnostic Test: 5-gene transcription signature — This is a prospective multisite diagnostic evaluation study to assess a novel approach to the diagnosis of enteric fever. The index test of host gene transcription responses by a 5 gene-signature will be compared to the reference test of blood culture confirmation for a diagnosis of enteric fever in patients with AUFI.

SUMMARY:
Acute undifferentiated febrile infection (AUFI) is a common presenting syndrome in low-resource settings and better diagnostics are urgently needed to improve patient management and guide disease prevention interventions. Assessment of the host gene expression response to infection in endemic populations has demonstrated significant promise as a new approach to identifying patients with enteric fever and for potential in differentiating between other causes of AUFI. Signatures identified through new data analytic techniques could be developed into a point-of-care test for use in endemic settings.

In this multisite diagnostic evaluation study we will collect prospective clinical, laboratory and diagnostic data from two endemic settings to evaluate host gene expression signatures for detecting enteric fever and for determining the cause of AUFI in LMIC settings.

ELIGIBILITY:
FEBRILE ADULTS- INCLUSION CRITERIA

* Age greater than or equal to 15 years and less than or equal to 65 years
* Participant is willing and they and/or an appropriate guardian/relative/representative is able to give informed consent for participation in the study and a follow-up (telephone) discussion at 14 days
* And either:

  1. Febrile illness without localising features (see 'exclusion criteria' and 'screening' sections) where fever is defined as:

     * documented tympanic/rectal temperature of ≥ 38°C or an axillary/oral temperature of ≥ 37.8°C, or a reported fever within the last 24 hours and
     * Reported duration of fever 3-14 days or
  2. Recently confirmed blood culture indicating enteric fever (confirmed within the previous 5 days)
* They may have had recent exposure to antimicrobials.

FEBRILE ADULTS- EXCLUSION CRITERIA

* The participant may not enter the study if ANY of the following apply:
* Unable to provide informed consent and no next of kin is willing and able to provide informed consent.
* For patients with febrile illness (included in (1) above): Any history or clinical suspicion of:

  * Rheumatological or connective tissue disorder (e.g. Rheumatoid arthritis)
  * Autoimmune condition (e.g. Autoimmune Hepatitis)
  * Malignancy
  * Active treatment with immunomodulating medications, or for tuberculosis (pulmonary or extrapulmonary) or any other chronic infection.
* Pregnancy (breast feeding mothers will NOT be excluded)
* No hospitalisation for more than 48 hours in the last 4 weeks
* Vaccination within 4 weeks prior to current admission
* Localising signs or symptoms of infection sufficient to diagnose the likely cause of acute febrile illness and thus prevent it from being 'undifferentiated.'

CONTROLS- INCLUSION CRITERIA

* Participant is willing and they are (and in 15-18 year olds, a guardian is) able to give informed consent for participation in the study
* Age greater than or equal to 15 years and less than or equal to 65 years
* They live outside of the normal/local catchment area for each hospital site
* Afebrile (as defined by no reported fever and temperature ≤ 38°C or an axillary/oral temperature of ≤ 37.8°C).

CONTROLS- EXCLUSION CRITERIA

* The participant may not enter the study if ANY of the following apply:
* Unable to provide informed consent and no next of kin (or parent/guardian in the case of a minor) is willing and able to provide informed consent.
* Current treatment for or prior history, or clinical suspicion of:

  * Rheumatological or connective tissue disorder
  * Autoimmune condition
  * Malignancy
  * Active treatment for tuberculosis (pulmonary or extrapulmonary) or clinical suspicion of active tuberculosis. Previous completed treatment is not a reason for exclusion.
  * Active treatment with immunomodulating medications or any other chronic infection.
* Pregnant (breast feeding mothers will NOT be excluded)
* Hospitalisation within 4 weeks of recruitment
* Vaccination within 4 weeks prior to recruitment
* Antimicrobial use within 4 weeks of recruitment
* Participant reports feeling more unwell than usual on the day of enrolment.

EXPLORATORY AIMS- PAEDIATRIC CRITERIA; INCLUSION CRITERIA

* Age greater than or equal to 2 years and less than 15 years
* As above for adult participants.

EXPLORATORY AIMS- PAEDIATRIC CRITERIA; EXCLUSION CRITERIA

* Parent/guardian is unwilling, and/or patient aged 8 to 14 years is unwilling to assent to provide informed consent.
* As above for adult participants.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We will recruit adults aged 15 to 65 years presenting to hospital with fever at 2 sites: 1 in Asia and 1 in Africa where enteric fever is endemic. All included febrile participants will have a (documented) tympanic/rectal temperature of ≥ 38°C or an axillary/oral temperature of ≥ 37.8°C on presentation and will report a history of fever within the last 24 hours lasting 3 to 14 days. In parallel, healthy community control participants will be recruited from each site catchment area during the course of the study with enrolment designed to result in an even representation of age groups and seasonal variation. Identified signatures of infection will be explored in a cohort of febrile children aged 2 to 14 years at each site. 600 febrile adults, 200 febrile children and 200 afebrile adult controls will be recruited at each site.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity (AUROC) of a diagnostic score derived from transcriptional responses by a 5-gene transcription signature (STAT1, SLAMF8, PSME2, WARS, ALDH1A1) in classifying patients with blood culture-confirmed enteric fever. | 2.5 years
  Evaluate the performance of a host gene transcription signature for detecting enteric fever in adults presenting with acute undifferentiated fever (AUFI)

SECONDARY OUTCOMES:
Number of participants with diagnosis confirmed by laboratory testing. | 2.5 years
  Determine the frequency of other common causes of AUFI at each site.
Number of participants presenting with mild, moderate or severe illness by clinical diagnosis according to validated prognostic scores such as sepsis scoring systems. | 2.5 years
  Assess the relationship between markers of clinical illness severity, likely infection cause and level of molecular perturbation.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Darton, Study Director — University of Sheffield
Locations (1):
- Christian Medical Centre, Vellore, India